CLINICAL TRIAL: NCT01504594
Title: Safeness and Effectiveness of Autologous Hematopoietic Cell Infusion Through Catheterization in Pediatric Patients With Dilated Cardiomyopathy
Brief Title: Autologous Stem Cells in Pediatric Patients With Dilated Cardiomyopathy
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Suspended because the lack of patients among the time this clinical trial was running.
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Consuelo Mancias Guerra, Pediatric Hematology Professor, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE-2012
Record Dates: First submitted 2011-12-15; First posted 2012-01-05 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Cardiomyopathy, Dilated
Keywords: Dilated cardiomyopathy; Idiopathic; Bone Marrow; Stem Cells; CD34 +; Autologous
MeSH Terms: conditions — Cardiomyopathy, Dilated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients (Experimental): Children which meet eligibility criteria and after being assessed, are stimulated with G-CSF, undergo bone marrow extraction and then have them applied directly to the coronary arteries through cardiac catheterization.
  Interventions: Procedure: Intracoronary autologous stem cell infusion

INTERVENTIONS:
Procedure: Intracoronary autologous stem cell infusion — Under sedation and under sterile conditions in a fluoroscopy operation room, cardiac catheterization will be performed through the femoral artery to infuse the stem cells directly into the heart´s coronary arteries.
  Other Names: Intracoronary CD34+ cell infusion

SUMMARY:
The purpose of this study is to determine whether an autologous stem cell infusion through catheterism is safe and effective in the treatment of pediatric dilated cardiomyopathy.

Process:

1. Primary Evaluation

   * Clinical History
   * Echocardiogram to evaluate ejection fraction and other parameters
2. Signing of Informed Consent and clearing doubts
3. Bone Marrow stimulation for 3 consecutive days with G-CSF (Granulocyte Colony Stimulating Factor) applied subcutaneously
4. On the 4th day, in operation room and under sedation: Bone Marrow Harvest performed by hematologists through posterior iliac crests(amount calculated at 8cc/kg, without exceeding 150ml).
5. Recovery room with family members while the cells are being processed in the Hematology Laboratory.
6. Approximately 3 hours after the 1st procedure, the patient re-enters the operation room, which is equipped for cardiac catheterization, so that cardiologists infuse the stem cells through the femoral artery into the coronary arteries which irrigate the heart´s muscle fibers.
7. Patient goes back to the recovery area until the anesthesia effect is gone and can tolerate oral liquids.
8. Clinical and echocardiographic follow-ups at 6 weeks and 6 months after the procedure.

DETAILED DESCRIPTION:
* The Patient will receive standard surgical care, accompanied by a nurse at all times.
* Premedication includes: Omeprazole (gastric protector), Ketorolac (anti-pain and swelling), ondansetron (antivomiting).

ELIGIBILITY:
Inclusion Criteria:

* Ejection fraction less than 35 percent in echocardiogram
* More than 3 months with complete medical treatment without significant improvement
* Complete medical treatment: digitalics, diuretics, vasodilators and beta blockers

Exclusion Criteria:

* Not signing informed consent
* Active infection at enrolling time
* Inadequate G-CSF application

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Safeness of autologous bone marrow derived stem cells infused through cardiac catheterization to coronary arteries. | 6 weeks
  Patient will be assessed to prove that the procedure did not cause any deterioration of his/her health presented at the beginning of the study.

SECONDARY OUTCOMES:
Effectiveness of autologous bone marrow derived stem cells infused through cardiac catheterization to coronary arteries. | 6 months
  Patient will be assessed to measure and record any possible changes in his/her clinical and echocardiographic studies that will reflect improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Consuelo Mancias, Hematologist, Study Director — Hematology Service, University Hospital of Monterrey; Gerardo Sanchez, Cardiologist, Principal Investigator — Pediatrics Service, University Hospital of Monterrey
Locations (1):
- University Hospital Dr. Jose E. Gonzalez, Monterrey, N.l., Mexico

REFERENCES:
- See also: University Hospital Dr. Jose E. Gonzalez — http://www.medicina.uanl.mx/hu/